CLINICAL TRIAL: NCT03770806
Title: Factors Affecting the Speed of Recovery After Anterior Cruciate Ligament Reconstruction
Brief Title: Factors Affecting the Speed of Recovery After ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Vanessa Loland, Associate Professor, Anesthesiology and Pain Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 51788
Record Dates: First submitted 2017-05-15; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Anterior Cruciate Ligament Injury; ACL Injury; ACL - Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: Subjects who choose to have medication alone with no block for their routine care will be in an observational group only with no randomization. Subjects who elect to have a nerve block placed for their routine treatment will be randomized per the research protocol to have the block placed at either the groin or the mid-thigh. Subjects in each study group will perform the same study procedures. This study will follow subjects for the first 6 months of their recovery to observe routine care pain treatments and evaluate whether the methods of pain control determine (a) severity and duration of postoperative pain, (b) the speed of recovery of muscle function, and (c) pain responses and aggressiveness of pursuing physical therapy maneuvers
Who Masked: Outcomes Assessor
Masking Description: The research coordinator in charge of checking in with subjects during the six month follow-up period is blind to the pain treatment condition of the subject (Groin block vs. Mid-thigh block
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Femoral Nerve Block (Experimental): Standard Ultrasound-guided femoral nerve block with Ropivacaine 0.5% and Dexamethasone 6-8mg. These subjects will also receive the standard multimodal oral premedication of Celebrex 300-400mg, Tylenol 1000mg, and Oxycontin 10mg.
  Interventions: Procedure: Femoral Nerve Block
- Adductor Canal Nerve Block (Experimental): Standard Ultrasound-guided adductor nerve block, mid-thigh, with Ropivacaine 0.5% and Dexamethasone 6-8mg. These subjects will also receive the standard multimodal oral premedication of Celebrex 300-400mg, Tylenol 1000mg, and Oxycontin 10mg.
  Interventions: Procedure: Adductor Nerve Block
- No Block (Experimental): For subjects who choose to have medication alone with no block for their routine care, there will be no changes to their care, which includes receiving the multimodal oral premedication of Celebrex 300-400mg, Tylenol 1000mg, and Oxycontin 10mg. They will be in an observational group only with no randomization.
  Interventions: Other: No Block

INTERVENTIONS:
Procedure: Femoral Nerve Block — Standard Ultrasound-guided peri-neural femoral nerve block with Ropivacaine 0.5% and Dexamethasone 6-8mg.
  Other Names: Oral preoperative Celebrex(celecoxib) 300-400 mg; Oral preoperative acetaminophen 1000 mg; Oral preoperative oxycontin (Oxycodone HCl) 10 mg
  Arms: Femoral Nerve Block
Procedure: Adductor Nerve Block — Standard Ultrasound-guided peri-neural adductor nerve block, mid-thigh, with Ropivacaine 0.5% and Dexamethasone 6-8mg
  Other Names: Oral preoperative Celebrex(celecoxib) 300-400 mg; Oral preoperative acetaminophen 1000 mg; Oral preoperative oxycontin (Oxycodone HCl) 10 mg
  Arms: Adductor Canal Nerve Block
Other: No Block — routine iv and oral pain medication alone-observation only
  Other Names: Oral preoperative Celebrex(celecoxib) 300-400 mg; Oral preoperative acetaminophen 1000 mg; Oral preoperative oxycontin (Oxycodone HCl) 10 mg
  Arms: No Block

SUMMARY:
The purpose of this study is to find out how postoperative pain affects recovery after anterior cruciate ligament (ACL) repair. Complete recovery after ACL repair involves healing of tissues at the surgical site, but also recovery of strength of the muscles that control movements at the knee. Some pain is normally experienced after ACL repair; the severity is variable from one individual to another. Pain is usually controlled by intravenous and oral (by mouth) pain medicines. It is also frequently controlled by numbing nerves that supply sensation to the knee joint and surrounding tissues. This procedure is called a nerve block.

The investigators want to determine if standard methods of pain control after surgery affect future pain control, and the ability to exercise and recover muscle strength after surgery. The investigators are also interested in determining what other factors, such as age, gender, anxiety, or coping skills might be predictive of pain severity and speed of recovery. As part of the study, the investigators will record subject's ratings of pain severity, use of painkiller medicines, and muscle bulk measured by standardized tests, at various time intervals in the first 6 months after surgery. The investigators will also ask them to complete two questionnaires,one that enquires about subject's responses to pain in the past (catastrophizing test), and one that measures anxiety they might have about surgery or pain on the day of surgery. The investigators will be studying approximately 180 people who are having ACL repair at University of Washington. Subjects may be involved who are having multiple ligaments repaired including the anterior cruciate ligament

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) tears of the knee are frequently repaired by surgically implanting a tendon graft in place of the torn original cruciate ligament. The graft may be taken from the patient having the repair (an autologous graft) or from a cadaver (an allograft). Complete recovery from surgical repair of an anterior cruciate ligament reconstruction requires that the graft becomes firmly engrafted at the site, surrounding tissues are healed and strength is restored in muscles that control movements at the knee. The recovery process typically requires from six months to one year. Pain in the early phase of recovery is typically moderate to severe and may be a major factor determining patient return to normal activity. It may also be a major factor limiting the patient's ability to cooperate with rehabilitation maneuvers.

Traditional methods of treatment for pain include use of opioid pain killers (such as morphine) and/or femoral nerve block at the groin. The potential hazards of opioid pain killers include opioid side effects (nausea, vomiting, constipation, drowsiness, respiratory depression and the potential for developing opioid dependency=addiction). Pain in the early phase of recovery, if severe, can lead to changes in the spinal cord that predispose to amplifying pain sensations, thus intensifying the need for pain killer medicines, a process referred to as "windup" or neuroplasticity. Similarly, the use of opioid pain killers may activate pain amplification systems potentially contributing to persistence of pain and favoring development of chronic pain. For these reasons, there is a belief that early aggressive efforts to treat postoperative pain, and minimize the use of opioid pain killers, can have significant benefits to patients both by improving their comfort level after surgery; facilitating rehabilitation efforts and return to normal activity.

Anesthesiologists at the University of Washington may use pain medicines alone and/or perform a nerve block to help patients undergoing ACL repair with their pain control. Patients are given a choice as to their desired methods of pain control. These options are normally discussed by the regional block team with the patient prior to surgery and the merits of each discussed. Approximately 60-70% of patients typically request the use of nerve blocks in the recovery unit to help control their pain. For those patients who choose a nerve block, the anesthesiologist will choose to perform the nerve block at the level of the groin or the mid thigh. This decision varies by provider and is typically random in nature. Both locations for the nerve block appear to work most of the time and each may have small differences: the speed of onset is typically faster when performed at groin level, while quadriceps muscle function may be less affected when performed at mid thigh. Neither method is known to be superior for this type of surgery. Because patients are non-weight bearing for at least the first 24 hours after surgery and must use crutches for mobilization, the weakening of the quadriceps muscles may be relatively unimportant during that time.

The investigators hypothesize that pain treatment after ACL reconstruction which includes a nerve block in combination with other pain medications will be associated with better pain control immediately after surgery and will minimize the need for patients to use opioid pain killers and experience common opioid- related side effects. A secondary hypothesis is that the effectiveness of pain control, whether by pain medicines, and/or in combination with nerve blocks will determine the patient's ability to perform routine activities of daily living in the acute phase (0-7 days), and subsequently may affect their ability to perform physical therapy maneuvers that are prescribed for their routine care.

STUDY PURPOSE

Aim 1: Determine whether pain reported by patients after surgery is related to the type of pain control utilized - (1) either intravenous and oral pain medication alone, (2) combined with nerve block at the groin, or (3) combined with nerve block at the mid thigh.

Aim 2: Examine whether pain severity affects the ability of patients to perform activities of daily living in the acute phase (recovery index measured at 7 days), and physical therapy maneuvers in the ensuing 6 months after surgery possibly retarding restoration of muscle function in the affected leg.

Aim 3: Determine whether preoperative psychologic tests designed to assess patients' coping skills (Pain Catastrophizing score) and anxiety (Stait anxiety index) predict postoperative pain reported by patients, acute phase recovery scores (recovery index), and rehabilitation endpoints

ELIGIBILITY:
INCLUSION Criteria:

* Subjects must be age 18-65,
* Subjects must be undergoing ACL repair at UWMC
* Subjects must be between an anesthesia risk category of 1-3
* Subjects must be candidates to have a nerve block if they should choose so.
* Subjects must be free of neurologic disease or coagulation defects
* Subjects must have no allergies to typical medications used during nerve blocks.
* Subjects must be fluent in English, able to read, and understand English readily in person or and/over the phone.

EXCLUSION Criteria:

* Any patients under 18 or over 75
* Patients with a BMI in excess of 40
* Non-English speaking patients
* Patients with allergies to nerve block medications
* Patients with neurological disease or coagulation defects
* Patients not undergoing ACL repair at UWMC
* Patients who are opioid tolerant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
Verbal Pain Scores | 30 minutes after block treatment
  self- reported verbal pain score where 0= no pain and 10 = worst imaginable
Verbal Pain Scores | while walking 24 hours after block treatment
  self- reported verbal pain score where 0= no pain and 10 = worst imaginable
Verbal Pain Scores | While walking 48 hours after block treatment
  self- reported verbal pain score where 0= no pain and 10 = worst imaginable
Verbal Pain Scores | While walking 7 days after block treatment
  self- reported verbal pain score where 0= no pain and 10 = worst imaginable
Verbal Pain Scores | While walking 2 weeks after block treatment
  self- reported verbal pain score where 0= no pain and 10 = worst imaginable
Verbal Pain Scores | While walking 4 weeks after block treatment
  self- reported verbal pain score where 0= no pain and 10 = worst imaginable
Verbal Pain Scores | While walking 2 months after block treatment
  self- reported verbal pain score where 0= no pain and 10 = worst imaginable
Verbal Pain Scores | While walking 3 months after block treatment
  self- reported verbal pain score where 0= no pain and 10 = worst imaginable
Verbal Pain Scores | While walking 4 months after block treatment
  self- reported verbal pain score where 0= no pain and 10 = worst imaginable
Verbal Pain Scores | While walking 5 months after block treatment
  self- reported verbal pain score where 0= no pain and 10 = worst imaginable
Verbal Pain Scores | While walking 6 months after block treatment
  self- reported verbal pain score where 0= no pain and 10 = worst imaginable

SECONDARY OUTCOMES:
Pain Catastrophizing Score | Pre-Operative measure-performed in preoperative holding area immediately before surgery
  The pain catastrophizing score " is a self-rating scale designed to measure the extent to which subjects have certain thoughts and feelings when they have experienced painful situations in the past . The goal is to identify the extent to which subjects magnify the effects of pain, ruminate about pain, or feel helpless in the face of pain, collectively described as "catastrophizing".. It consists of 13 questions rated 0- 4 in response to the Prefix "When I'm in Pain, I worry….. with 0 being not at all, and 4 being all the time. The maximum total score is 52 Maximum score of 52 would indicate severe catastrophizing tendency, and 0 none. The results of 3 subscales are summed (magnification , rumination and helplessness ) for the final score.where 0= not a catastrophizer, and 52 would be the greatest level of catastrophizing about pain
Abbreviated State Anxiety Score | Pre-Operative Measure-performed in preopertive holding area immediately before surgery
  This scale is designed to assesses patients' state of anxiety preoperatively on the day of surgery.. A questionnaire that is a validated short form of the State-Trait anxiety test is used .
  It consists of 6 questions relating to the patient's current state of anxiety. It is administered in the preoperative holding area before the subjects have they receive any medication. They are asked how they feel on a scale of 1-4 with 1-being not at all, and 4 being very much so, in response to being asked if they feel Calm, tense, upset, relaxed, content or worried. The scores for positive (non- anxious) emotions are reversed numerically to convert high numbers to low numbers, and the anxious responses remain positive with the highest numbers (4) indicating the highest level of anxiety. The results of the converted 6 components are then summed.
  The maximum anxiety score is 24 = very anxious; the minimum is 0 = not anxious at all
Physical Therapy milestones-duration of activity | At physical therapy appointment 4 weeks after block treatment
  Minutes of rehab exercises/week time spent doing physical therapy exercises/week
Physical Therapy milestones-mobility | At physical therapy appointment 4 weeks after block treatment
  Degrees of knee flexion and extension, thigh circumference in each leg
Physical Therapy milestones-duration of activity | At physical therapy appointment 2 months after block treatment
  Minutes of rehab exercises/week
Physical Therapy milestones-mobility | At physical therapy appointment 2 months after block treatment
  Degrees of knee flexion and extension, thigh circumference in each leg
Physical Therapy milestones-duration of activity | At physical therapy appointment 3 months after block treatment
  Minutes of rehab exercises/week
Physical Therapy milestones-mobility | At physical therapy appointment 3 months after block treatment
  Degrees of knee flexion and extension, thigh circumference in each leg
Physical Therapy milestones-duration of activity | At physical therapy appointment 4 months after block treatment
  Minutes of rehab exercises/week
Physical Therapy milestones-mobility | At physical therapy appointment 4 months after block treatment
  Degrees of knee flexion and extension, thigh circumference in each leg
Physical Therapy milestones-duration of activity | At physical therapy appointment 5 months after block treatment
  Minutes of rehab exercises/week
Physical Therapy milestones-mobility | At physical therapy appointment 5 months after block treatment
  Degrees of knee flexion and extension, thigh circumference in each leg
Physical Therapy milestones-duration of activity | At physical therapy appointment 6 months after block treatment
  Minutes of rehab exercises/week
Physical Therapy milestones-mobility | At physical therapy appointment 6 months after block treatment
  Degrees of knee flexion and extension, thigh circumference in each leg
Self-reported Verbal Pain scores correlational analysis | 24 hours after block treatment
  correlate verbal pain scores with opioid use at 0-24 hrs (Spearmans correlation coefficient)
Self-reported Verbal Pain scores correlational analysis | 48 hours after block treatment
  correlate verbal pain scores with opioid use at 24-48hrs (Spearman'scorrelation coefficient)
Self-reported Verbal Pain scores correlational analysis | 7 days after block treatment
  Correlate recovery index with verbal pain scores (Pearson, and spearman's r)
Self-reported Verbal Pain scores correlational analysis | 2 weeks after block treatment
  correlate verbal pain scores with knee flexion and extension, and duration of exercise (Spearman's r)
Self-reported Verbal Pain scores correlational analysis | 4 weeks after block treatment
  correlate verbal pain scores with knee flexion and extension, and duration of exercise (Spearman's r)
Self-reported Verbal Pain scores correlational analysis | 2 months after block treatment
  correlate verbal pain scores with knee flexion and extension and duration of exercise (Spearman's r)
Self-reported Verbal Pain scores | 3 months after block treatment
  correlate verbal pain scores with knee flexion and extension and duration of exercise (Spearman's r)
Self-reported Verbal Pain scores | 4 months after block treatment
  correlate verbal pain scores with knee flexion and extension and duration of exercise (Spearman's r)
Self-reported Verbal Pain scores | 5 months after block treatment
  correlate verbal pain scores with knee flexion and extension and duration of exercise (Spearman's r)
Self-reported Verbal Pain scores | 6 months after block treatment
  correlate verbal pain scores with knee flexion and extension and duration of exercise (Spearman's r)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreae MH, Andreae DA. Regional anaesthesia to prevent chronic pain after surgery: a Cochrane systematic review and meta-analysis. Br J Anaesth. 2013 Nov;111(5):711-20. doi: 10.1093/bja/aet213. Epub 2013 Jun 28. PMID 23811426
- [Background] Ong CK, Lirk P, Seymour RA, Jenkins BJ. The efficacy of preemptive analgesia for acute postoperative pain management: a meta-analysis. Anesth Analg. 2005 Mar;100(3):757-773. doi: 10.1213/01.ANE.0000144428.98767.0E. PMID 15728066
- [Background] Grevstad U, Mathiesen O, Valentiner LS, Jaeger P, Hilsted KL, Dahl JB. Effect of adductor canal block versus femoral nerve block on quadriceps strength, mobilization, and pain after total knee arthroplasty: a randomized, blinded study. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):3-10. doi: 10.1097/AAP.0000000000000169. PMID 25376972
- [Background] Sawyer S. Femoral nerve block for pain relief after total knee replacement. Prof Nurse. 2004 Feb;19(6):333-7. PMID 14983606
- [Background] Johnson RL, Duncan CM, Ahn KS, Schroeder DR, Horlocker TT, Kopp SL. Fall-prevention strategies and patient characteristics that impact fall rates after total knee arthroplasty. Anesth Analg. 2014 Nov;119(5):1113-8. doi: 10.1213/ANE.0000000000000438. PMID 25211392
- [Background] Hanson NA, Allen CJ, Hostetter LS, Nagy R, Derby RE, Slee AE, Arslan A, Auyong DB. Continuous ultrasound-guided adductor canal block for total knee arthroplasty: a randomized, double-blind trial. Anesth Analg. 2014 Jun;118(6):1370-7. doi: 10.1213/ANE.0000000000000197. PMID 24842182
- [Background] Williams BA, Kentor ML, Vogt MT, Irrgang JJ, Bottegal MT, West RV, Harner CD, Fu FH, Williams JP. Reduction of verbal pain scores after anterior cruciate ligament reconstruction with 2-day continuous femoral nerve block: a randomized clinical trial. Anesthesiology. 2006 Feb;104(2):315-27. doi: 10.1097/00000542-200602000-00018. PMID 16436852
- [Background] Ilfeld BM, Meyer RS, Le LT, Mariano ER, Williams BA, Vandenborne K, Duncan PW, Sessler DI, Enneking FK, Shuster JJ, Maldonado RC, Gearen PF. Health-related quality of life after tricompartment knee arthroplasty with and without an extended-duration continuous femoral nerve block: a prospective, 1-year follow-up of a randomized, triple-masked, placebo-controlled study. Anesth Analg. 2009 Apr;108(4):1320-5. doi: 10.1213/ane.0b013e3181964937. PMID 19299806
- [Background] Kwofie MK, Shastri UD, Gadsden JC, Sinha SK, Abrams JH, Xu D, Salviz EA. The effects of ultrasound-guided adductor canal block versus femoral nerve block on quadriceps strength and fall risk: a blinded, randomized trial of volunteers. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):321-5. doi: 10.1097/AAP.0b013e318295df80. PMID 23788068
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Pavlin DJ, Sullivan MJ, Freund PR, Roesen K. Catastrophizing: a risk factor for postsurgical pain. Clin J Pain. 2005 Jan-Feb;21(1):83-90. doi: 10.1097/00002508-200501000-00010. PMID 15599135
- [Background] Hart DL, Werneke MW, George SZ, Matheson JW, Wang YC, Cook KF, Mioduski JE, Choi SW. Screening for elevated levels of fear-avoidance beliefs regarding work or physical activities in people receiving outpatient therapy. Phys Ther. 2009 Aug;89(8):770-85. doi: 10.2522/ptj.20080227. Epub 2009 Jun 18. PMID 19541772
- [Background] Asmundson GJ, Bovell CV, Carleton RN, McWilliams LA. The Fear of Pain Questionnaire-Short Form (FPQ-SF): factorial validity and psychometric properties. Pain. 2008 Jan;134(1-2):51-8. doi: 10.1016/j.pain.2007.03.033. Epub 2007 May 4. PMID 17482361
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159
- [Background] Csintalan RP, Inacio MC, Funahashi TT. Incidence rate of anterior cruciate ligament reconstructions. Perm J. 2008 Summer;12(3):17-21. doi: 10.7812/TPP/07-140. PMID 21331205
- [Background] Luo TD, Ashraf A, Dahm DL, Stuart MJ, McIntosh AL. Femoral nerve block is associated with persistent strength deficits at 6 months after anterior cruciate ligament reconstruction in pediatric and adolescent patients. Am J Sports Med. 2015 Feb;43(2):331-6. doi: 10.1177/0363546514559823. Epub 2014 Dec 2. PMID 25466410
- [Background] Krych A, Arutyunyan G, Kuzma S, Levy B, Dahm D, Stuart M. Adverse effect of femoral nerve blockade on quadriceps strength and function after ACL reconstruction. J Knee Surg. 2015 Feb;28(1):83-8. doi: 10.1055/s-0034-1371769. Epub 2014 Mar 12. PMID 24622910
- [Background] Peters ML, Sommer M, de Rijke JM, Kessels F, Heineman E, Patijn J, Marcus MA, Vlaeyen JW, van Kleef M. Somatic and psychologic predictors of long-term unfavorable outcome after surgical intervention. Ann Surg. 2007 Mar;245(3):487-94. doi: 10.1097/01.sla.0000245495.79781.65. PMID 17435557
- [Background] Wong J, Tong D, De Silva Y, Abrishami A, Chung F. Development of the functional recovery index for ambulatory surgery and anesthesia. Anesthesiology. 2009 Mar;110(3):596-602. doi: 10.1097/ALN.0b013e318197a16d. PMID 19212260